CLINICAL TRIAL: NCT01542502
Title: Pilot Feasibility Study of the Safety and Efficacy of Anakinra in Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM14079
Record Dates: First submitted 2012-02-23; First posted 2012-03-02 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Heart Failure
Keywords: Heart failure with preserved ejection fraction; Diastolic heart failure; Aerobic exercise performance
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Experimental): Treatment with daily subcutaneous injections of Anakinra 100 mg
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Treatment with daily subcutaneous injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Anakinra 100 mg daily subcutaneous injection
  Other Names: Recombinant human Interleukin-1 receptor antagonist; Kineret
  Arms: Anakinra
Drug: Placebo — Placebo daily subcutaneous injection
  Other Names: Sodium Chloride (NaCl) 0.9%
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, crossover pilot study to measure the safety and feasibility of Interleukin-1 (IL-1) blockade with Anakinra in patients with stable heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of congestive heart failure
* Recent Imaging Study (<12 months) showing Left Ventricular Ejection Fraction (LVEF) >50% and Left Ventricular End Diastolic Volume Index (LVEDVI) <97ml/m2
* Evidence of abnormal Left Ventricular (LV) relaxation, filling, diastolic distensibility, and diastolic stiffness as shown by one of the following:

  1. Invasive Hemodynamic measurements

     * mean Pulmonary Capillary Wedge pressure (mPCW) >12
     * Left Ventricular End Diastolic Pressure (LVEDP) >16 mmHg
  2. Tissue Doppler Echocardiogram

     * E/E' >15
     * E/E' 8-15 and one of the following

       * Left Ventricular Hypertrophy (LVH)
       * Atrial Fibrillation
       * Left Atrial Enlargement
       * E/A <0.5 + Deceleration Time (DT) >280 (if >50yrs of age)
  3. Biomarkers
* Brain Natriuretic Peptide (BNP) >200pg/mL

Exclusion Criteria:

* Age <18
* Recent changes (previous 3 months) in HF maintenance medications (beta-blockers, angiotensin converting enzyme [ACE] inhibitors, aldosterone antagonists, vasodilators, cardiac glycosides, diuretics)
* Hospitalization for worsening Heart Failure (HF) or acute decompensated HF within the previous 12months
* Anticipated need for cardiac resynchronization therapy (CRT) or automated-implantable cardioverter defibrillator (AICD)
* Angina or electrocardiograph (ECG) changes that limit maximum exertion during cardiopulmonary exercise testing
* Active infection including chronic infection
* Active cancer
* Recent (<14 days) use of anti-inflammatory drugs (not including Non-Steroidal Anti-Inflammatory Drugs [NSAIDs]), Chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus), malignancy, or any comorbidity limiting survival or ability to complete the study
* Pregnancy (determined by urine pregnancy test in women of childbearing potential)
* Inability to give informed consent
* Other conditions limiting completion of cardiopulmonary exercise test or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anakinra (First) Then Placebo (Second): Treatment with daily subcutaneous injections of Anakinra 100 mg for 14 days, followed by daily subcutaneous injections of Placebo for 14 days
  Anakinra: Anakinra 100 mg daily subcutaneous injection Placebo: Placebo daily subcutaneous injection
- Placebo (First) Then Anakinra (Second): Treatment with daily subcutaneous injections of Placebo for 14 days, followed by daily subcutaneous injections of Anakinra for 14 days
  Placebo: Placebo daily subcutaneous injection Anakinra: Anakinra 100 mg daily subcutaneous injection
Period: Overall Study
Arm/Group | Anakinra (First) Then Placebo (Second) | Placebo (First) Then Anakinra (Second)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a cross-over trial, so all patients have been treated with anakinra and with placebo at different times.
Groups:
- All Participants: Baseline measures for all study participants
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [55 to 64]
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Consumption (Peak VO2)
Description: The primary endpoint is the change in peak oxygen consumption among stable heart failure patients (n = 12) following 14-days treatment with daily doses of Anakinra 100 mg (SC, subcutaneous).
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: ml*kg^-1*min^-1
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 12 | 12
ml*kg^-1*min^-1 | 1.1 [0.6 to 2.3] | -0.1 [-0.5 to 1.0]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p = 0.009, ANOVA

2. Secondary Outcome: Exercise Time
Description: Interval change from baseline in duration of exercise during a standardized cardiopulmonary exercise test upon completion of 2 weeks treatment
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Anakinra: Treatment with daily subcutaneous injections of Anakinra
  Anakinra: Anakinra 100 mg daily subcutaneous injection
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 12 | 12
minutes | 0.05 [-0.05 to 0.85] | 0.4 [0.025 to 0.925]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p = 0.87, ANOVA

3. Other Pre Specified Outcome: Correlation Between Endpoints
Description: Correlation between interval change in peak VO2 and high sensitivity C-reactive protein
Time Frame: 28 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Heart Failure Symptoms (DASI)
Description: Interval change from baseline in Heart Failure (HF) symptoms as measured by Duke Activity Status Index (DASI) upon completion of 2 weeks treatment.
Time Frame: 28 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Adverse Events
Description: Additional endpoints will include assessment of adverse events and hospitalizations during 4-week duration of study.
Time Frame: 28 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Inflammatory Biomarkers
Description: Interval change from baseline in high-sensitivity C-reactive protein upon completion of 2 weeks treatment.
Time Frame: 28 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Ventilatory Efficiency (VE/VCO2 [Carbon Dioxide] Slope)
Description: Interval change from baseline in ventilatory efficiency (VE/VCO2 slope) upon completion of 2 weeks treatment.
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Anakinra | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=12) | Placebo (N=12)
Injection site reactions (Skin and subcutaneous tissue disorders) | 3 | 0 — Mild injection site reaction - not requiring cessation of therapy

LIMITATIONS AND CAVEATS:
This is a pilot study to estimate the effects of targeted anti-inflammatory treatment on aerobic exercise capacity in patients with Heart Failure and Preserved Ejection Fraction. All findings should therefore be considered hypothesis generating.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes